CLINICAL TRIAL: NCT01552486
Title: Biology and Clinical Outcomes of Chiropractic Spinal Manipulative Therapy in the Treatment of Patients With Acute Inflammatory Radiculopathy Secondary to Lumbar Disc Herniation: a Pilot Study
Brief Title: Chiropractic Spinal Manipulative Therapy for Acute Sciatica Secondary to Lumbar Disc Herniation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Vancouver General Hospital (Other)
Responsible Party: Principal Investigator, Dr. Paul Bishop, Clinical Associate Professor, I.C.O.R.D. Research Professor, Division of Spine, Department of Orthopaedics, University of British Columbia, Vancouver General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 1R21AT006773-01A1 (NIH)
Record Dates: First submitted 2012-02-29; First posted 2012-03-13 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Acute Sciatica; Lumbar Disc Herniation
Keywords: chiropractic; manipulation; radiculopathy; sciatica; lumbar; disc; herniation; protrusion
MeSH Terms: conditions — Intervertebral Disc Displacement; Radiculopathy; Sciatica; Hernia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chiropractic Spinal Manipulative Therapy (Experimental)
  Interventions: Other: Chiropractic Spinal Manipulative Therapy
- Usual Care (Other)
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Chiropractic Spinal Manipulative Therapy — Patients will receive a course high-velocity low-amplitude thrust spinal manipulation 3 times per week for 4 weeks.
  Arms: Chiropractic Spinal Manipulative Therapy
Other: Usual Care — Patients will be under the care of the their general physician and will be allowed the following medications: gabapentin, pregabalin, nortriptyline, amitriptyline.
  Arms: Usual Care

SUMMARY:
Comparisons of surgical and non-operative treatment of patients with acute sciatica secondary to lumbar intervertebral disc herniation (AS/LDH) have shown no appreciable difference in outcome. The composition of the non-operative treatment of this patient population remains poorly defined. Spinal manipulative therapy (SMT) has demonstrated value in the treatment of AS/LDH. Recent preliminary studies suggest that SMT provides therapeutic benefit through the modulation of in vivo inflammatory mediators. This feasibility study will define the key experimental variables required to conduct a large multicentre study that will clarify the biological and clinical outcomes of SMT in the treatment of patients with AS/LDH.

ELIGIBILITY:
Inclusion Criteria:

* chief complaint of sciatica rather than lower back pain
* pain of up to 6 months' duration
* a McCulloch criteria score of 5/5 (two clinical symptoms and two clinical signs of sciatica, and diagnostic imaging confirming the presence of a herniated nucleus pulposus contacting a spinal nerve root at the appropriate level)
* fluency in spoken and written English to ensure subjects understand the content of questionnaires and consent

Exclusion Criteria:

* progressive neurological deficit
* spinal fracture
* spinal tumor
* spinal infection
* spinal nerve root motor score of less than 4/5
* spinal stenosis that is not attributable to a herniated disc
* any other significant spinal ailment or local or generalized co-morbidity ailment that could affect outcomes independently of SMT ( e.g. seronegative spondyloarthropathy, malignancy).

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Rate of recruitment of eligible patients | The number of patients recruited per week for 19 months

SECONDARY OUTCOMES:
Cytokine and cytokine mRNA levels in serum. | Change from baseline cytokine and cytokine mRNA levels in serum 4 weeks prior to surgery or commencing chiropractic spinal manipulative therapy (CSMT).
Cytokine and cytokine mRNA levels in serum | Change from baseline cytokine and mRNA levels in serum pre-surgery or following a 4-week course of CSMT.
Cytokine and cytokine mRNA levels in serum | Change from baseline cytokine and mRNA levels in serum and 12 weeks post-surgery and/or post-CSMT
Cytokine and cytokine mRNA levels in serum. | Change from baseline cytokine and mRNA levels in serum and 24 weeks post-surgery and/or post-CSMT
Total mRNA levels (isolated from disc tissue and disc / periradicular lavage samples) of interleukins 1,10 and 11, MIP-1 beta TNF alpha, and chemotactic protein alpha. | Specimens will be harvested an average of 6 weeks post-randomization
Modified Roland Disability Questionnaire (mRDQ) score and Visual Analogue Scale (VAS) pain scale. | Change from baseline and 4-weeks prior to surgery or commencing 4-weeks of CSMT.
mRDQ and VAS | Change from baseline and pre-surgery or following a 4-week course of CSMT
mRMQ and VAS | Change from baseline and 12 weeks post-surgery and/or post-CSMT
mRDQ and VAS | Change from baseline and 24 weeks post-surgery and/or post-CSMT

CONTACTS AND LOCATIONS:
Overall Officials: Paul B Bishop, DC, MD, PhD, Principal Investigator — Clinical Associate Professor, I.C.O.R.D. Research Professor, Division of Spine, Department of Orthopaedics, University of British Columbia
Locations (1):
- Integrated Spine Clinic, Blusson Spinal Cord Centre, Vancouver General Hospital, Vancouver, British Columbia, Canada